CLINICAL TRIAL: NCT00233324
Title: Surfactant Positive Airway Pressure and Pulse Oximetry Trial (SUPPORT) in Extremely Low Birth Weight Infants
Brief Title: Surfactant Positive Airway Pressure and Pulse Oximetry Trial
Acronym: SUPPORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Neonatal Research Network (Network)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: NICHD-NRN-0033; U10HD021364 (NIH); U10HD021373 (NIH); U10HD021385 (NIH); U10HD027851 (NIH); U10HD027853 (NIH); U10HD027856 (NIH); U10HD027871 (NIH); U10HD027880 (NIH); U10HD027904 (NIH); U10HD034216 (NIH); U10HD036790 (NIH); U10HD040461 (NIH); U10HD040492 (NIH); U10HD040689 (NIH); U10HD053089 (NIH); U10HD053109 (NIH); U10HD053119 (NIH); U10HD053124 (NIH); UL1RR024128 (NIH); UL1RR024139 (NIH); UL1RR024979 (NIH); UL1RR024982 (NIH); UL1RR024989 (NIH); UL1RR025008 (NIH); M01RR000633 (NIH); M01RR000750 (NIH); M01RR008084 (NIH); U10HD021397 (NIH); U10HD040521 (NIH); U10HD040498 (NIH)
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Results first posted 2014-12-05 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Infant, Newborn, Diseases; Other Preterm Infants; Infant, Small for Gestational Age; Premature Birth; Bronchopulmonary Dysplasia; Retinopathy of Prematurity
Keywords: NICHD Neonatal Research Network; Extremely Low Birth Weight (ELBW); Very Low Birth Weight (VLBW); Prematurity; Mechanical ventilation; Surfactant; Intubation; Neurodevelopmental impairment; Pulse oximetry; Oxygen saturation; Positive-Pressure Respiration
MeSH Terms: conditions — Infant, Newborn, Diseases; Premature Birth; Bronchopulmonary Dysplasia; Retinopathy of Prematurity | interventions — Surface-Active Agents; Continuous Positive Airway Pressure; high-potential iron-sulfur protein oxygen oxidoreductase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Surfactant and Low Oxygen (Experimental): Administration of surfactant by endotracheal tube and supplemental oxygen with target saturation of 85% to 89%
  Interventions: Drug: Surfactant; Drug: Supplemental oxygen with target saturation of 85 to 89%
- Surfactant and High Oxygen (Experimental): Administration of surfactant by endotracheal tube and supplemental oxygen with target saturationof 91% to 95%
  Interventions: Drug: Surfactant; Drug: Supplemental oxygen with target saturation of 91 to 95%
- CPAP and Low Oxygen (Experimental): Administration of continuous positive airway pressure (CPAP) and supplemental oxygen with target saturation of 85% to 89%
  Interventions: Device: Continuous Positive Airway Pressure (CPAP); Drug: Supplemental oxygen with target saturation of 85 to 89%
- CPAP and High Oxygen (Experimental): Administration of continuous positive airway pressure (CPAP)and supplemental oxygen with target saturation of 91% to 95%
  Interventions: Device: Continuous Positive Airway Pressure (CPAP); Drug: Supplemental oxygen with target saturation of 91 to 95%

INTERVENTIONS:
Drug: Surfactant — Intubation and administration of surfactant by 1 hour of age.
  Arms: Surfactant and High Oxygen; Surfactant and Low Oxygen
Device: Continuous Positive Airway Pressure (CPAP) — Continuous Positive Airway Pressure/Positive End Expiratory Pressure (CPAP/PEEP) begun in the delivery room and continuing in the NICU
  Other Names: CPAP
  Arms: CPAP and High Oxygen; CPAP and Low Oxygen
Drug: Supplemental oxygen with target saturation of 85 to 89% — Supplemental oxygen in the range of 85% to 89% until the infant is no longer requiring ventilatory support or oxygen
  Other Names: Low oxygen
  Arms: CPAP and Low Oxygen; Surfactant and Low Oxygen
Drug: Supplemental oxygen with target saturation of 91 to 95% — Supplemental oxygen in the range of 91% to 95% until the infant is no longer requiring ventilatory support or oxygen.
  Other Names: High oxygen
  Arms: CPAP and High Oxygen; Surfactant and High Oxygen

SUMMARY:
This study compared the use of continuous positive airway pressure initiated at birth with the early administration of surfactant administered through a tube in the windpipe within 1 hour of birth for premature infants born at 24 to 27 weeks gestation. In addition, these infants within 2 hours of birth, had a special pulse oximeter placed to continuously monitor their oxygen saturation in two different target ranges (85-89% or 91-95%). This study helped determine whether or not these two management strategies affect chronic lung disease and survival of premature infants.

DETAILED DESCRIPTION:
Study subjects were infants of 24 0/7ths to 27 6/7th weeks at birth for which a decision has been made to provide full resuscitation as required. Infants 27 weeks or less gestation (completed weeks by best obstetric estimate) were enrolled because more than 80% of such infants in the Network are intubated, usually early in their neonatal course. The feasibility trial demonstrated that the five NICHD centers involved could reduce intubation in the delivery room to less than 50% of such infants if they are not intubated for surfactant. We excluded infants of 23 weeks or less in view of their extremely high mortality and morbidity, and their almost universal need for delivery room intubation for resuscitation. Secondary studies included: neuroimaging/MRI, growth, and breathing outcomes.

Strata: There were two randomization strata, infants of 24 0/7ths to 25 6/7ths weeks, and infants of 26 0/7ths-27 6/7ths weeks by best obstetrical estimate.

Randomization:

Randomization was stratified by gestational age group, occurred prior to delivery for consented deliveries, and was performed by utilizing specially prepared double-sealed envelopes. Deliveries were randomized as a unit, thus multiples, twins, triplets, etc. were randomized to the same arm of the trial.

Informed Consent:

Parents were approached prior to delivery for informed consent, and their infants enrolled at delivery.

Study Intervention: Mode of Ventilatory Support The intervention began after birth when the infant was given to the resuscitation team. The conduct of the resuscitation followed usual guidelines, and once stabilized, all Control infants in both strata received prophylactic/early surfactant (within one hour of age), whereas all Treatment infants were placed on CPAP/PEEP following stabilization, and were intubated only for resuscitation indications.

Pulse Oximeter Allocation:

Infants were randomized to receive either a high- or low-saturation of peripheral oxygen (SpO2) as monitored by a study oximeter immediately following NICU admission, with a maximum allowable delay of two hours following admission.

The SUPPORT Trial recruitment was temporarily paused on November 23, 2005 based on concern regarding pulse oximeter readings > 95% and due to concern regarding separation of the two arms of the oximetry portion of the study. Further analyses were performed which showed that infants on room air accounted for a significant portion of pulse oximetry saturations above 95%. Separation of the two groups was reanalyzed based on time spent in room air and the duration of time spent at individual SpO2 values, which both showed group differences. The trial was restarted on February 6, 2006.

Follow-up: Subjects will be seen for a follow-up visit at 18-22 months corrected age to look at neurodevelopment.

Extended follow-up: Subjects enrolled in the Neuroimaging/MRI secondary study will also be seen for a follow-up visit at 6-7 years to look at later school-age development. Subjects attending the 6-7 year follow-up visit will be invited to participate in this secondary study which will analyze the relationship of salivary cortisol and dehydroepiandrosterone (DHEA) to: (a) blood pressure and adiposity; (b) prenatal and postnatal growth; and (c) DNA methylation patterns.

ELIGIBILITY:
Inclusion Criteria:

* Infants with a minimal gestational age of 24 weeks 0 days to 27 completed weeks (up to 27 6/7ths) by best obstetrical estimate
* Infants who will receive full resuscitation as necessary, i.e., no parental request or physician decision to forego resuscitation
* Infants whose parents/legal guardians have provided consent for enrollment, or
* Infants without known major congenital malformations

Exclusion Criteria:

* Any infant transported to the center after delivery
* Infants whose parents/legal guardians refuse consent
* Infants born during a time when the research apparatus/study personnel are not available
* Infants < 24 weeks 0 days or > 28 weeks 0 days, completed weeks of gestation

Ages: 24 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1316 (Actual)
Dates: Start 2005-02; Primary Completion 2009-02 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abbot R. Laptook, MD, Principal Investigator — Brown University, Women & Infants Hospital of Rhode Island; Michele C. Walsh, MD MS, Principal Investigator — Case Western Reserve University, Rainbow Babies and Children's Hospital; Ronald N. Goldberg, MD, Principal Investigator — Duke University; Barbara J. Stoll, MD, Principal Investigator — Emory University; Brenda B. Poindexter, MD MS, Principal Investigator — Indiana University; Abhik Das, PhD, Principal Investigator — RTI International; Krisa P. Van Meurs, MD, Principal Investigator — Stanford University; Ivan D. Frantz III, MD, Principal Investigator — Tufts Medical Center; Neil N. Finer, MD, Principal Investigator — University of California, San Diego; Kurt Schibler, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Waldemar A. Carlo, MD, Principal Investigator — University of Alabama at Birmingham; Edward F. Bell, MD, Principal Investigator — University of Iowa; Kristi L. Watterberg, MD, Principal Investigator — University of New Mexico; Pablo J. Sanchez, MD, Principal Investigator — University of Texas, Southwestern Medical Center at Dallas; Kathleen A. Kennedy, MD MPH, Principal Investigator — The University of Texas Health Science Center, Houston; Roger G. Faix, MD, Principal Investigator — University of Utah; Seetha Shankaran, MD, Principal Investigator — Wayne State University; Richard A. Ehrenkranz, MD, Principal Investigator — Yale University
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Tufts Medical Center, Boston, Massachusetts
  - Wayne State University, Detroit, Michigan
  - University of New Mexico, Albuquerque, New Mexico
  - University of Rochester, Rochester, New York
  - Wake Forest University, Charlotte, North Carolina
  - RTI International, Durham, North Carolina
  - Duke University, Durham, North Carolina
  - Cincinnati Children's Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Brown University, Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Deuticke B. Monocarboxylate transport in red blood cells: kinetics and chemical modification. Methods Enzymol. 1989;173:300-29. doi: 10.1016/s0076-6879(89)73020-2. No abstract available. PMID 2674614
- [Result] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Carlo WA, Finer NN, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Schibler K, Newman NS, Ambalavanan N, Frantz ID 3rd, Piazza AJ, Sanchez PJ, Morris BH, Laroia N, Phelps DL, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Ehrenkranz RA, Watterberg KL, Higgins RD. Target ranges of oxygen saturation in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1959-69. doi: 10.1056/NEJMoa0911781. Epub 2010 May 16. PMID 20472937
- [Result] SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network; Finer NN, Carlo WA, Walsh MC, Rich W, Gantz MG, Laptook AR, Yoder BA, Faix RG, Das A, Poole WK, Donovan EF, Newman NS, Ambalavanan N, Frantz ID 3rd, Buchter S, Sanchez PJ, Kennedy KA, Laroia N, Poindexter BB, Cotten CM, Van Meurs KP, Duara S, Narendran V, Sood BG, O'Shea TM, Bell EF, Bhandari V, Watterberg KL, Higgins RD. Early CPAP versus surfactant in extremely preterm infants. N Engl J Med. 2010 May 27;362(21):1970-9. doi: 10.1056/NEJMoa0911783. Epub 2010 May 16. PMID 20472939
- [Result] Rich WD, Auten KJ, Gantz MG, Hale EC, Hensman AM, Newman NS, Finer NN; National Institute of Child Health and Human Development Neonatal Research Network. Antenatal consent in the SUPPORT trial: challenges, costs, and representative enrollment. Pediatrics. 2010 Jul;126(1):e215-21. doi: 10.1542/peds.2009-3353. Epub 2010 Jun 29. PMID 20587676
- [Result] Di Fiore JM, Walsh M, Wrage L, Rich W, Finer N, Carlo WA, Martin RJ; SUPPORT Study Group of Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Low oxygen saturation target range is associated with increased incidence of intermittent hypoxemia. J Pediatr. 2012 Dec;161(6):1047-52. doi: 10.1016/j.jpeds.2012.05.046. Epub 2012 Jun 26. PMID 22738947
- [Result] Rich W, Finer NN, Gantz MG, Newman NS, Hensman AM, Hale EC, Auten KJ, Schibler K, Faix RG, Laptook AR, Yoder BA, Das A, Shankaran S; SUPPORT and Generic Database Subcommittees of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Enrollment of extremely low birth weight infants in a clinical research study may not be representative. Pediatrics. 2012 Mar;129(3):480-4. doi: 10.1542/peds.2011-2121. Epub 2012 Feb 27. PMID 22371462
- [Result] Ambalavanan N, Carlo WA, Wrage LA, Das A, Laughon M, Cotten CM, Kennedy KA, Laptook AR, Shankaran S, Walsh MC, Higgins RD; SUPPORT Study Group of the NICHD Neonatal Research Network. PaCO2 in surfactant, positive pressure, and oxygenation randomised trial (SUPPORT). Arch Dis Child Fetal Neonatal Ed. 2015 Mar;100(2):F145-9. doi: 10.1136/archdischild-2014-306802. Epub 2014 Nov 25. PMID 25425651
- [Result] Navarrete CT, Wrage LA, Carlo WA, Walsh MC, Rich W, Gantz MG, Das A, Schibler K, Newman NS, Piazza AJ, Poindexter BB, Shankaran S, Sanchez PJ, Morris BH, Frantz ID 3rd, Van Meurs KP, Cotten CM, Ehrenkranz RA, Bell EF, Watterberg KL, Higgins RD, Duara S; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Growth Outcomes of Preterm Infants Exposed to Different Oxygen Saturation Target Ranges from Birth. J Pediatr. 2016 Sep;176:62-68.e4. doi: 10.1016/j.jpeds.2016.05.070. Epub 2016 Jun 22. PMID 27344218
- [Result] Stevens TP, Finer NN, Carlo WA, Szilagyi PG, Phelps DL, Walsh MC, Gantz MG, Laptook AR, Yoder BA, Faix RG, Newman JE, Das A, Do BT, Schibler K, Rich W, Newman NS, Ehrenkranz RA, Peralta-Carcelen M, Vohr BR, Wilson-Costello DE, Yolton K, Heyne RJ, Evans PW, Vaucher YE, Adams-Chapman I, McGowan EC, Bodnar A, Pappas A, Hintz SR, Acarregui MJ, Fuller J, Goldstein RF, Bauer CR, O'Shea TM, Myers GJ, Higgins RD; SUPPORT Study Group of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Respiratory outcomes of the surfactant positive pressure and oximetry randomized trial (SUPPORT). J Pediatr. 2014 Aug;165(2):240-249.e4. doi: 10.1016/j.jpeds.2014.02.054. Epub 2014 Apr 13. PMID 24725582
- [Result] Vaucher YE, Peralta-Carcelen M, Finer NN, Carlo WA, Gantz MG, Walsh MC, Laptook AR, Yoder BA, Faix RG, Das A, Schibler K, Rich W, Newman NS, Vohr BR, Yolton K, Heyne RJ, Wilson-Costello DE, Evans PW, Goldstein RF, Acarregui MJ, Adams-Chapman I, Pappas A, Hintz SR, Poindexter B, Dusick AM, McGowan EC, Ehrenkranz RA, Bodnar A, Bauer CR, Fuller J, O'Shea TM, Myers GJ, Higgins RD; SUPPORT Study Group of the Eunice Kennedy Shriver NICHD Neonatal Research Network. Neurodevelopmental outcomes in the early CPAP and pulse oximetry trial. N Engl J Med. 2012 Dec 27;367(26):2495-504. doi: 10.1056/NEJMoa1208506. PMID 23268664
- [Derived] Lowe J, Bann CM, Dempsey AG, Fuller J, Taylor HG, Gustafson KE, Watson VE, Vohr BR, Das A, Shankaran S, Yolton K, Ball MB, Hintz SR; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Do Bayley-III Composite Scores at 18-22 Months Corrected Age Predict Full-Scale IQ at 6-7 Years in Children Born Extremely Preterm? J Pediatr. 2023 Dec;263:113700. doi: 10.1016/j.jpeds.2023.113700. Epub 2023 Aug 26. PMID 37640232
- [Derived] Lowe J, Fuller JF, Dempsey AG, Do B, Bann CM, Das A, Gustafson KE, Vohr BR, Hintz SR, Watterberg KL; SUPPORT NEURO School-Age Study Subcommittee of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Cortisol awakening response and developmental outcomes at 6-7 years in children born extremely preterm. Pediatr Res. 2023 Feb;93(3):689-695. doi: 10.1038/s41390-022-02113-9. Epub 2022 Jun 17. PMID 35715492
- [Derived] Duncan AF, Bann CM, Dempsey AG, Adams-Chapman I, Heyne R, Hintz SR; Eunice Kennedy Shriver National Institute of Child Health and Development Neonatal Research Network. Neuroimaging and Bayley-III correlates of early hand function in extremely preterm children. J Perinatol. 2019 Mar;39(3):488-496. doi: 10.1038/s41372-019-0314-0. Epub 2019 Jan 28. PMID 30692613
- [Derived] Duncan AF, Bann CM, Dempsey A, Peralta-Carcelen M, Hintz S; Eunice Kennedy Shriver National Institute of Child Health and Development Neonatal Research Network. Behavioral Deficits at 18-22 Months of Age Are Associated with Early Cerebellar Injury and Cognitive and Language Performance in Children Born Extremely Preterm. J Pediatr. 2019 Jan;204:148-156.e4. doi: 10.1016/j.jpeds.2018.08.059. Epub 2018 Oct 3. PMID 30292492
- [Derived] Chawla S, Natarajan G, Shankaran S, Carper B, Brion LP, Keszler M, Carlo WA, Ambalavanan N, Gantz MG, Das A, Finer N, Goldberg RN, Cotten CM, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Markers of Successful Extubation in Extremely Preterm Infants, and Morbidity After Failed Extubation. J Pediatr. 2017 Oct;189:113-119.e2. doi: 10.1016/j.jpeds.2017.04.050. Epub 2017 Jun 7. PMID 28600154
- [Derived] Di Fiore JM, Martin RJ, Li H, Morris N, Carlo WA, Finer N, Walsh M; SUPPORT Study Group of the Eunice Kennedy Shriver National Institute of Child Health, and Human Development Neonatal Research Network. Patterns of Oxygenation, Mortality, and Growth Status in the Surfactant Positive Pressure and Oxygen Trial Cohort. J Pediatr. 2017 Jul;186:49-56.e1. doi: 10.1016/j.jpeds.2017.01.057. Epub 2017 Mar 6. PMID 28279433
- [Derived] Hintz SR, Barnes PD, Bulas D, Slovis TL, Finer NN, Wrage LA, Das A, Tyson JE, Stevenson DK, Carlo WA, Walsh MC, Laptook AR, Yoder BA, Van Meurs KP, Faix RG, Rich W, Newman NS, Cheng H, Heyne RJ, Vohr BR, Acarregui MJ, Vaucher YE, Pappas A, Peralta-Carcelen M, Wilson-Costello DE, Evans PW, Goldstein RF, Myers GJ, Poindexter BB, McGowan EC, Adams-Chapman I, Fuller J, Higgins RD; SUPPORT Study Group of the Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neuroimaging and neurodevelopmental outcome in extremely preterm infants. Pediatrics. 2015 Jan;135(1):e32-42. doi: 10.1542/peds.2014-0898. Epub 2014 Dec 1. PMID 25554820
- [Derived] LeVan JM, Brion LP, Wrage LA, Gantz MG, Wyckoff MH, Sanchez PJ, Heyne R, Jaleel M, Finer NN, Carlo WA, Das A, Stoll BJ, Higgins RD; Eunice Kennedy Shriver NICHD Neonatal Research Network. Change in practice after the Surfactant, Positive Pressure and Oxygenation Randomised Trial. Arch Dis Child Fetal Neonatal Ed. 2014 Sep;99(5):F386-90. doi: 10.1136/archdischild-2014-306057. Epub 2014 May 29. PMID 24876196
- See also: NICHD Neonatal Research Network site — http://neonatal.rti.org/
- See also: NICHD Pregnancy & Perinatology Branch — https://www.nichd.nih.gov/about/org/der/branches/ppb/Pages/projects.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3546 infants assessed for eligibility from 3127 pregnancies. 2230 were excluded for not meeting eligibility criteria or parental permission was not granted or other reasons.
Pre-assignment Details: 235 did not meet eligiblity criteria 125 did not have personnel or equipment available 699 were eligible did not have consent sought 344 were eligible but parent or guardian was not available 748 were eligible but parent or guardian denied permission to enroll 68 were eligible and had permission but were not randomized 11 had other reasons
Groups:
- Early Surfactant and Lower Range Oxygen: Early Surfactant and 85-89% target oxygen saturation
- Early Surfactant and Higher Range Oxygen: Early Surfactant and 91-95% target oxygen saturation
- CPAP and Lower Range Oxygen: Continuous Positive Airway Pressure (CPAP) and 85-89% target oxygen saturation
- CPAP and Higher Range Oxygen: Continuous Positive Airway Pressure (CPAP) and 91-95% target oxygen saturation
Period: Main Study
Arm/Group | Early Surfactant and Lower Range Oxygen | Early Surfactant and Higher Range Oxygen | CPAP and Lower Range Oxygen | CPAP and Higher Range Oxygen
Started | 318 | 335 | 336 | 327
Completed | 250 | 275 | 274 | 280
Not Completed | 68 | 60 | 62 | 47
Not completed — Death | 68 | 60 | 62 | 47
Period: Follow up at 18-22 Months Corrected Age
Arm/Group | Early Surfactant and Lower Range Oxygen | Early Surfactant and Higher Range Oxygen | CPAP and Lower Range Oxygen | CPAP and Higher Range Oxygen
Started | 250 | 275 | 274 | 280
Completed | 237 | 261 | 256 | 269
Not Completed | 13 | 14 | 18 | 11
Not completed — Death | 5 | 7 | 5 | 4
Not completed — Undetermined retinopathy status | 8 | 7 | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- CPAP and Lower Range Oxygen: Continuous Positive Airway Pressure/Positive End Expiratory Pressure (CPAP/PEEP) begun in the delivery room and continuing in the NICU and oxygen administered in lower range (85-90%)
- CPAP and Higher Range Oxygen: Continuous Positive Airway Pressure/Positive End Expiratory Pressure (CPAP/PEEP) begun in the delivery room and continuing in the NICU and oxygen adminstered in higher range (91-95%)
- Early Surfactant and Lower Range Oxygen: Intubation and administration of surfactant by 1 hour of age and oxygen adminstered in lower range (85-90%)
- Early Surfactant and Higher Range Oxygen: Intubation and administration of surfactant by 1 hour of age and oxygen adminstered in higher range (91-95%)
- Total: Total of all reporting groups
Arm/Group | CPAP and Lower Range Oxygen | CPAP and Higher Range Oxygen | Early Surfactant and Lower Range Oxygen | Early Surfactant and Higher Range Oxygen | Total
Number analyzed (Participants) | 336 | 327 | 318 | 335 | 1316
Age, Customized [Number; unit: participants]
  >23 weeks and <28 weeks gestational age | 336 | 327 | 318 | 335 | 1316
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 149 | 141 | 142 | 604
  Male | 164 | 178 | 177 | 193 | 712
Region of Enrollment [Number; unit: participants]
  United States | 336 | 327 | 318 | 335 | 1316

OUTCOME MEASURES:

1. Primary Outcome: Survival Without Bronchopulmonary Dysplasia (BPD)
Time Frame: 36 weeks
Measure: Number; unit: Participants
Groups:
- CPAP: Continuous Positive Airway Pressure/Positive End Expiratory Pressure (CPAP/PEEP) begun in the delivery room and continuing in the NICU
Arm/Group | CPAP | Surfactant
Number analyzed (Participants) | 663 | 653
Participants | 346 | 320

2. Primary Outcome: Survival Without Severe Retinopathy of Prematurity (ROP) (Threshold Disease or the Need for Surgery)
Time Frame: 55 weeks
Population: 49 infants in the lower oxygen saturation group and 46 infants in the higher oxygen saturation group that had unknown retinopathy of prematurity outcome
Measure: Number; unit: participants
Groups:
- Lower Oxygen Saturation Target: SpO2 range (85% to 89%) until the infant is no longer requiring ventilatory support or oxygen.
- Higher Oxygen Saturation Target: SpO2 range (91% to 95%) until the infant is no longer requiring ventilatory support or oxygen.
Arm/Group | Lower Oxygen Saturation Target | Higher Oxygen Saturation Target
Number analyzed (Participants) | 605 | 616
participants | 434 | 418

3. Secondary Outcome: Death or Neurodevelopmental Impairment
Time Frame: 18-22 months
Measure: Number; unit: participants
Arm/Group | CPAP | Surfactant | Lower Oxygen Saturation Target | Higher Oxygen Saturation Target
Number analyzed (Participants) | 621 | 613 | 612 | 622
participants | 173 | 183 | 185 | 171

4. Secondary Outcome: Duration of Mechanical Ventilation
Description: The length in days that an individual was on mechanical ventilation which includes high frequency and conventional ventilation.
Time Frame: Entire NICU stay, up to 120 days
Population: 1078 participants survived to discharge and they all had information available for regarding use of mechanical ventilation.
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Surfactant and High Oxygen: Administration of surfactant by endotracheal tube and supplemental oxygen with target saturation of 91% to 95%
- CPAP and High Oxygen: Administration of continuous positive airway pressure (CPAP) and supplemental oxygen with target saturation of 91% to 95%
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 249 | 275 | 274 | 280
days | 11 [2 to 32] | 13 [2 to 37] | 7 [1 to 29] | 11.5 [2 to 32.5]

5. Secondary Outcome: Survival Without Ventilation
Description: Surviving the first 7 days of life without any need for ventilation by day 7
Time Frame: From birth through first 7 days of life.
Population: 1307 participants had known survival and ventilation statuses. 9 participants were excluded due to unknown ventilation status from birth through 7 days of life: 6 infants in the lower oxygen group, 3 infants in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 317 | 335 | 331 | 324
Participants | 161 | 157 | 190 | 172

6. Secondary Outcome: Received Surfactant Treatment
Description: Received any surfactant treatment.
Time Frame: From birth through 120 days of life.
Population: 1312 participants had known surfactant treatment. 4 were excluded due to unknown surfactant treatment: 2 infants in the low oxygen group, 2 infants in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 317 | 335 | 335 | 325
Participants | 159 | 176 | 42 | 51

7. Secondary Outcome: Number of Participants With Air Leaks
Description: Number of participants with air leaks including pnemothorax, pulmonary interstitial emphysema (PIE), and pneumopericardium.
Time Frame: From birth through first 14 days of life.
Population: All 1316 participants had data on incidence of air leaks.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 318 | 335 | 336 | 327
Participants | 26 | 22 | 25 | 20

8. Secondary Outcome: Physiological Bronchopulmonary Dysplasia
Description: Infants who received support via ventilator or CPAP at 36 weeks PMA. Alternatively, infants who received low levels of supplemental oxygen (<30%) at 36 weeks PMA may have been eligible for a physiologic challenge in which there was an attempt to wean the infant to room air. Specifically, infants were eligible for the challenge if at 36 weeks PMA if they were receiving effective oxygen <27% and had majority saturation >90%, or they were receiving effective oxygen 27-30% and had majority saturation >96%, or they were receiving room air by nasal cannula. The challenge took place between 36 and 37 weeks PMA. Those who were not challenged because their level of support increased (support with CPAP or ventilation or increased oxygen) were considered to have BPD, as were those who failed the challenge.
Time Frame: 36 weeks post menstrual age.
Population: 1108 participants survived to 36 weeks and had BPD information. 208 participants did not survive to 36 weeks and were excluded: 114 from the low oxygen group, 94 from the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 258 | 281 | 282 | 287
Participants | 102 | 117 | 103 | 120

9. Secondary Outcome: Death
Description: Participants who died by their follow-up visit at 18-22 months.
Time Frame: 18-22 months
Population: 1281 participants with confirmed deaths or survivals by follow-up. 35 were excluded due to incomplete follow-up visits: 21 in low oxygen group, 14 in high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 310 | 328 | 323 | 320
Participants | 73 | 67 | 67 | 51

10. Secondary Outcome: Severe Intraventricular Hemorrhage (IVH)
Description: There are four grades of intraventricular hemorrhage: Grade I - echodensity/hemorrhage is confied to the germinal matrix. Grade II - echodensity/hemorrhage in the lateral ventricle(s) without distention. Grade III - echodensity/hemorrhage in the lateral ventricle(s) with distention. Grade IV - echodense lesion in the parenchyma. Severe IVH is defined as having IVH grades of III or IV.
Time Frame: From birth through first 120 days of life.
Population: 1270 participants had known IVH grades. 46 were excluded due to unknown IVH status: 24 infants from the low oxygen group, 22 infants from high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 307 | 321 | 323 | 319
Participants | 34 | 38 | 49 | 43

11. Secondary Outcome: Periventricular Leukomalacia (PVL)
Description: Increased echogenicity or cysts in periventricular region.
Time Frame: From birth through first 120 days of life.
Population: 1272 participants had known PVL statuses. 44 were excluded due to unknown PVL status: 23 infants in the low oxygen group, 21 infants in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 307 | 322 | 324 | 319
Participants | 10 | 16 | 14 | 14

12. Secondary Outcome: Threshold Retinopathy of Prematurity (ROP) Requiring Surgery
Description: Diagnosis of retinopathy of prematurity which resulted in requiring surgery.
Time Frame: From birth through first 120 days of life.
Population: 997 surviving participants with ROP data were included. 319 total participants were excluded due to death (N=224) or missing ROP data (N=95): 171 in the low oxygen group, 148 in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 230 | 250 | 253 | 264
Participants | 19 | 44 | 17 | 47

13. Secondary Outcome: Endotracheal Intubation
Description: Insertion of a tube into the trachea to allow positive pressure ventilation for breathing.
Time Frame: Delivery Room, post-delivery
Population: 1312 participants had non-missing data on whether they experienced endotracheal intubation. 4 participants were excluded due to missing information: 2 infants in the low oxygen group, 2 infants in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 317 | 335 | 335 | 325
Participants | 294 | 315 | 110 | 117

14. Secondary Outcome: Duration of Oxygen Supplementation
Description: The length of time in days that a participant had oxygen supplementation.
Time Frame: From birth through first 120 days of life.
Population: 1078 participants survived to discharge and they all had information available regarding the duration of their oxygen supplementation.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 249 | 275 | 274 | 280
days | 46 [21 to 87] | 60 [33 to 93] | 43 [15 to 71] | 59 [28.5 to 88]

15. Secondary Outcome: Pulse Oximetry Values > 90%
Description: Percentage of time spent above 90% oxygen saturation.
Time Frame: From birth through first 120 days of life.
Population: 90 were excluded due to incomplete data: 48 from the low oxygen saturation group and 42 from the high oxygen saturation group.
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 302 | 314 | 304 | 306
percentage of time | 62 [53 to 73] | 76 [70 to 81] | 63 [55 to 73] | 77 [71 to 83]

16. Secondary Outcome: Blindness in at Least One Eye
Description: Blindness in at least one eye by 18-22 months of life.
Time Frame: 18-22 months
Population: 990 participants survived and were seen at the 18-22 month follow-up. 326 were excluded: 175 in the low oxygen group, 151 in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 225 | 254 | 254 | 257
Participants | 4 | 3 | 1 | 5

17. Secondary Outcome: Received Postnatal Steroids
Description: Participant received any doses or courses of systemic steroids to prevent or treat bronchopulmonary dysplasia/chronic lung disease.
Time Frame: From birth through first 120 days of life.
Population: 1280 participants had information regarding whether they received postnatal steroids. 36 participants were excluded due to missing data: 18 infants in the low oxygen group, 18 infants in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 308 | 323 | 328 | 321
Participants | 42 | 41 | 19 | 28

18. Secondary Outcome: Necrotizing Enterocolitis (NEC)
Description: Proven necrotizing enterocolitis (NEC) diagnosis using the Modified Bell's Staging Criteria for NEC.
Time Frame: From birth through first 120 days of life.
Population: 1290 participants had known NEC statuses. 26 were excluded due to missing NEC data: 13 infants in the low oxygen group, 13 infants in the high oxygen group.
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 311 | 325 | 330 | 324
Participants | 36 | 27 | 40 | 43

19. Secondary Outcome: Cerebral Palsy
Description: Incidence of cerebral palsy.
Time Frame: 18-22 months
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 225 | 254 | 254 | 257
Participants | 17 | 17 | 26 | 24

20. Other Pre Specified Outcome: Apgar Scores at 5 Minutes
Description: Apgar stands for "Appearance, Pulse, Grimace, Activity, and Respiration" and scores range from 1 (worst) to 10 (best) indicating a baby's condition 5 minutes after birth.
Time Frame: 5 minutes after birth.
Population: All 1316 participants had APGAR scores at 5 minutes.
Measure: Median (Inter-Quartile Range); unit: scores on a scale
Arm/Group | Surfactant and Low Oxygen | Surfactant and High Oxygen | CPAP and Low Oxygen | CPAP and High Oxygen
Number analyzed (Participants) | 318 | 335 | 336 | 327
scores on a scale | 7 [6 to 8] | 7 [6 to 8] | 7 [6 to 8] | 7 [6 to 8]

ADVERSE EVENTS:
Groups:
- Surfactant and Lower Range Oxygen: Early Surfactant and 85-89% target oxygen saturation
- Surfactant and Higher Range Oxygen: Early Surfactant and 91-95% target oxygen saturation
Arm/Group | Surfactant and Lower Range Oxygen | Surfactant and Higher Range Oxygen | CPAP and Lower Range Oxygen | CPAP and Higher Range Oxygen
Serious Adverse Events (participants affected / at risk) | 204/318 | 227/335 | 231/336 | 224/327
Other Adverse Events (participants affected / at risk) | 4/318 | 5/335 | 11/336 | 7/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Surfactant and Lower Range Oxygen (N=318) | Surfactant and Higher Range Oxygen (N=335) | CPAP and Lower Range Oxygen (N=336) | CPAP and Higher Range Oxygen (N=327)
Death (General disorders) | 68 | 60 | 62 | 47
Chest compressions or drugs in the delivery room (Cardiac disorders) | 22 | 24 | 19/333 | 17 — Number at risk is lower than total entered on this arm due to missing data because of early death or other reasons.
Air leak during initial 14 days (Respiratory, thoracic and mediastinal disorders) | 26 | 22 | 25 | 20
Intraventricular hemorrhage (IVH) Grade 3 or 4 (Nervous system disorders) | 34/307 | 38/321 | 49/323 | 43/319 — Number at risk is lower than total entered on this arm due to study withdrawal of some participants due to death or other reasons.
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 24/311 | 21/325 | 20/330 | 13/324 — Number at risk is lower than total entered on this arm due to study withdrawal of some participants due to death or other reasons.
Necrotizing enterocolitis (Gastrointestinal disorders) | 36/311 | 27/325 | 40/330 | 43/324 — Number at risk is lower than total entered on this arm due to study withdrawal of some participants due to death or other reasons.
Patent Ductus Aretriosus (Cardiac disorders) | 151/311 | 160/325 | 156/330 | 164/323 — Number at risk is lower than total entered on this arm due to study withdrawal of some participants due to death or other reasons.
Nasal Breakdown (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Surfactant and Lower Range Oxygen (N=318) | Surfactant and Higher Range Oxygen (N=335) | CPAP and Lower Range Oxygen (N=336) | CPAP and Higher Range Oxygen (N=327)
Nasal Breakdown (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 10 | 6
Any other non-serious adverse event (General disorders) | 0 | 2 | 1 | 1 — Additional adverse events are available only at the summary level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No